CLINICAL TRIAL: NCT06539455
Title: Analysis of Liver Injury Risk Factors in a Multiethnic Population Treated With Antituberculosis Drugs
Acronym: TUBILI
Status: Active, not recruiting | Type: Observational
Sponsor: Stefania Cheli (Other)
Responsible Party: Sponsor-Investigator, Stefania Cheli, Study coordinator, ASST Fatebenefratelli Sacco
Organization: ASST Fatebenefratelli Sacco (Other)
Other Study IDs: TUBILI
Record Dates: First submitted 2024-07-30; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Tuberculosis Infection
Keywords: isoniazide; rifampicin; drug-induced injury liver (DILI); slow acetylator; genotyping
MeSH Terms: conditions — Latent Tuberculosis; Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Human DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- DILI group: Anti-TB DILI was defined by: 1) AST or ALT level > 5 times the ULN in patients with the absence of symptoms or with a total BIL level > 2 times the ULN; or 2) AST or ALT level > 3 times the ULN and total BIL level > 3 times the ULN in patients who show symptoms compatible with hepatitis.
  Interventions: Drug: standard anti-TB treatment
- Non-DILI group: Subjects who had no hepatotoxicity events during the therapeutic regimen
  Interventions: Drug: standard anti-TB treatment

INTERVENTIONS:
Drug: standard anti-TB treatment — standard anti-TB treatment in line with international guidelines (isoniazid , rifampin, ethambutol, and pyrazinamide)

SUMMARY:
Tuberculosis (TB) is the world's second leading cause of death from a single infectious agent after COVID-19. In 2022, TB was estimated to have affected 10.6 million people, of whom 1.3 million died because of it, despite the WHO's implementation of the "End TB" program. Although the gold standard therapy is effective, it may lead to adverse events, among which hepatotoxicity is the most common. Due to its frequency, severity, and potential outcome, anti-TB drug-induced liver injury (DILI) is extremely concerning. Despite decades of use and the large number of patients exposed to anti-TB drugs worldwide, the pathogenesis underlying DILI remains poorly understood. Investigation of drug-related, host genetic, and environmental factors associated with hepatotoxicity susceptibility, as well as studies examining potential mechanisms causing DILI, may help clinicians develop strategies for reducing the incidence of hepatotoxicity. The aim of this study was to determine host- and drug-related risk factors and their association with hepatotoxicity in a multiethnic population in order to enable early identification of individuals with increased susceptibility to anti-TB DILI. An improved understanding of these factors may help to predict and prevent the occurrence of DILI and develop more effective treatments.

DETAILED DESCRIPTION:
Tuberculosis (TB) is the world's second leading cause of death from a single infectious agent in 2022, after COVID-19. In 2022, TB disease was estimated to affect 10.6 million people, of whom 1.3 million died because of it, despite the WHO's adoption of the End TB Strategy. The standardised therapy involves a treatment regimen of isoniazid (INH), rifampin (RIF), ethambutol (EMB), and pyrazinamide (PZA) for 2 months, then INH and RMP for at least an additional 4-7 months [3]. Even though 85% of TB cases are successfully treated, significant morbidity from treatment-related adverse events, such as hepatotoxicity, skin reactions, and gastrointestinal and neurological disorders, reduces the efficacy of therapy. In 11% of patients receiving INH, RMP, and PZA in combination, hepatotoxicity is the most frequent adverse effect that results in drug discontinuation. One of the most prevalent subtypes of idiosyncratic hepatotoxicity is caused by anti-TB drugs. There are many factors contributing to the development of liver injury that are related both to the drug and to the patient's characteristics. As to drug-related factors, acetylhydrazine, which is generated by NAT2, is widely considered a crucial INH metabolite that contributes to drug-induced liver injury (DILI). Given the importance of acetylation in INH metabolism, several studies have investigated NAT2 loss of function polymorphisms as possible risk factors for anti-TB DILI. In addition, advanced age, female gender, poor nutritional status, HBV or HCV infection, HIV infection, chronic liver disease, and alcoholism are environmental, physiological, and pathological factors contributing to anti-TB DILI incidence. Geographic and ethnic characteristics also play a role in the occurrence of DILI. This event is also ascribed to the polymorphisms observed at the level of genes encoding for metabolic enzymes. Of note, most studies available in the literature have been conducted in Asiatic geographical areas, where TB is considered of great concern due to its high incidence. Moreover, it is well known that the Chinese population is commonly composed of NAT2 rapid acetylators, showing a lower susceptibility to the development of anti-TB DILI. There is still considerable controversy and uncertainty regarding the potential role that the acetylator status of individuals (rapid or slow) may play in INH-induced hepatotoxicity, given the fact that the results of previous studies have shown such considerable variability.

Due to the impossibility of treating liver injury, the only recovery strategy is drug discontinuation in tuberculosis patients; its prevention is essential to avoiding this condition. To prevent the progression of the disease, increase the efficiency of treatment, and reduce mortality, screening patients for risk factors may be extremely useful. Consequently, the current study's aim is to determine the association between anti-TB DILI incidence and potential environmental, physiologic, and pathologic factors. Since 2020, a cohort of patients has been followed in the Department of Infectious Diseases of Luigi Sacco Hospital in Milan, Italy. Moreover, despite the multi-ethnic characterisation of the cohort enrolled in this study, the high prevalence of Caucasian patients (who also present a greater frequency of slow acetylators) may be provide a complementary perspective to previously published studies, mostly focusing on Asian populations. Based on this cohort, we performed a nested case-control study to understand the role of several drug- and host-related factors in DILI.

ELIGIBILITY:
Inclusion criteria:

1. adult patients (>18 years)
2. patient who received standard initial therapy including INH (5mg/kg), RMP (10mg/kg), and PZA (25mg/kg) for patients with active TB disease
3. treatment with first line anti-TB drugs, including rifampicin and isoniazid for patients with latent TBI
4. normal serum ALT and bilirubin levels, no symptoms related to abnormal liver function prior to anti-TB drug treatment
5. informed consent.

Exclusion criteria:

1. liver dysfunction, including biliary origin, before anti-TB therapy
2. patients receiving non-standard treatment regimen initially (e.g., patients with severe pulmonary or extrapulmonary TB receiving large doses or more than four anti-TB drugs), 3) modified treatment regimen due to drug resistance or intolerance excluding first line anti-TB drugs

4) lactation or pregnancy 5) concomitant use of hepatotoxic drugs 6) abnormal hepatic function on laboratory testing before anti-TB 7) disease that was resistant to INH at the start of treatment 8) patients refusing to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data collected from patients with confirmed tuberculosis, enrolled at the Department of Infectious Diseases of Luigi Sacco Hospital in Milan, Italy, between July 2020 and September 2023, will be analysed. Subjects were all followed up as outpatients at Tuberculosis Clinic at Luigi Sacco Hospital, some of them with previous inward stays at various hospitals in the Lombardy Region.
  The participants were given standard anti-TB treatment in line with international guidelines (RMP 10 mg/kg, INH 5 mg/kg), primarily administered orally, although intravenous administration was employed for inpatients as needed, and modified to oral administration as soon as possible. The other drugs of the standard regimen included standard daily doses of PZA (15-30 mg/kg) and EMB (15-20 mg/kg).
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The occurrence of anti-TB DILI (number of participants with DILI) | 6-12 month
  Association between risk factors (drug- and host-related factors) and the incidence of DILI.
  Evaluation of patient characteristics associated with the development of DILI. DILI was defined by: 1) AST or ALT level > 5 times the ULN in patients with absence of symptoms or with total BIL level > 2 times the ULN, or 2) AST or ALT level > 3 time the ULN and total BIL level > 3 times the ULN in patients who show symptoms compatible with hepatitis.

SECONDARY OUTCOMES:
The prevalence of early hepatotoxicity experience | 6-12 month
  Evaluate the characteristics of patients who first experienced anti-TB DILI.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Fatebenefratelli Sacco, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheli S, Torre A, Schiuma M, Montrasio C, Civati A, Galimberti M, Battini V, Mariani I, Mosini G, Carnovale C, Radice S, Clementi E, Gori A, Antinori S. NAT2 Slow Acetylator Phenotype as a Significant Risk Factor for Hepatotoxicity Caused by Antituberculosis Drugs: Results From a Multiethnic Nested Case-Control Study. Clin Infect Dis. 2025 Aug 1;81(1):145-152. doi: 10.1093/cid/ciae583. PMID 39727196

DOCUMENTS (1):
  • Study Protocol (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT06539455/Prot_000.pdf